CLINICAL TRIAL: NCT06258434
Title: Liquid Biopsy Based Multiomics Study for the Detection of Colorectal Advanced Neoplasia in High Risk Chinese Patients: an Prospective, Single Bind Observational Study (COLO-LIMULOID)
Brief Title: Liquid Biopsy Based Multiomics Study for Colorectal Cancer Early Screening
Acronym: COLO-LIMULOID
Status: Not yet recruiting | Type: Observational
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Sheng Dai, Principal Investigator, head of medical affairs, Sir Run Run Shaw Hospital
Other Study IDs: 20211204-31
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer; Adenomatous Polyps; Adenoma; Advanced Adenoma
MeSH Terms: conditions — Colorectal Neoplasms; Adenomatous Polyps; Adenoma | interventions — Early Detection of Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — blood and stool sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high risk CRC screening group: Prospective enrollment of subjects with pre-defined high risk factors for developing colorectal cancer or CRC patients
  Interventions: Diagnostic Test: multiomics Colorectal Cancer (CRC) screening test (CRC-Appareo)
- CRC group: Prospective enrollment of subjects with confirmed colorectal cancer
  Interventions: Diagnostic Test: multiomics Colorectal Cancer (CRC) screening test (CRC-Appareo)

INTERVENTIONS:
Diagnostic Test: multiomics Colorectal Cancer (CRC) screening test (CRC-Appareo) — Patients who are at high risk of developing CRC or confirmed CRC and willing to conduct colonoscopy examination will be asked to collect blood prior to bowl preparation for multiomics CRC screening test which using Reduced Representation Bisulfite Sequencing (RRBS) technology to obtain multidimensional variation information on cell-free DNA (cfDNA) methylation, end sequence, fragment size distribution, and copy number variation in the blood, and integrate analysis through machine learning algorithms to accurately assess the risk of colorectal cancer and advanced adenoma. and will be asked to collect stool sample for commercially available FIT assay. Colonoscopy and histopathologic examination are used as reference. The diagnosis information of each sample was blind to the participants who conduct the multiomics profiling, as well as the informatics who perform the integrate analysis.
  Other Names: fecal immunochemical test（FIT ）; diagnostic colonoscopy

SUMMARY:
The primary objective is to determine the diagnostic sensitivity and specificity of the newly developed liquid biopsy based multiomics Colorectal Cancer (CRC) screening test (CRC-Appareo) for detecting advanced neoplasia (including colorectal cancer and advanced adenomas) in high risk patients and patients with confirmed CRC, using colonoscopy as the reference method. The secondary objective is to compare the screening performance of the multiomics Colorectal Cancer (CRC) screening test with commercially available FIT (Fecal Immunochemical Test) assay in detecting advanced neoplasia.

DETAILED DESCRIPTION:
The study will be carried out in 5 hospitals throughout China. Patients who are at high risk of developing CRC or confirmed CRC and willing to conduct colonoscopy examination will be asked to collect blood prior to bowl preparation for multiomics CRC screening test which using Reduced Representation Bisulfite Sequencing (RRBS) technology to obtain multidimensional variation information on cell-free DNA (cfDNA) methylation, end sequence, fragment size distribution, and copy number variation in the blood, and integrate analysis through machine learning algorithms to accurately assess the risk of colorectal cancer and advanced adenoma. and will be asked to collect stool sample for commercially available FIT assay. Colonoscopy and histopathologic examination are used as reference. The diagnosis information of each sample was blind to the participants who conduct the multiomics profiling, as well as the informatics who perform the integrate analysis.

ELIGIBILITY:
Inclusion Criteria:

Willing to provide written consent Able to provide blood and stool samples

For high risk CRC screening group:

Scheduled for colonoscopy voluntarily or by physician prescription

CRC high risk profile as defined below:

History of FIT positivity Family history of CRC Any of two of the following clinical symptoms: chronic constipation/diarrhea, stool with mucous, chronic appendicitis, chronic bilary track diseases, mental stress

For CRC group:

Confirmed CRC patients No prior treatment with chemotherapy, radiotherapy, and prior to any surgical procedures

Exclusion Criteria:

Unwilling to provide blood samples FAP (familial adenomatous polyposis), Crohn's disease, ulcerative colitis Prior history of colonoscopy within the past 5 years and removal of lesions History of CRC other conditions deemed not suited for the study by investigators

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with high risk of developing CRC and CRC patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-02-10 (Estimated); Primary Completion 2024-08-10 (Estimated); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the multiomics Colorectal Cancer (CRC) screening test (CRC-Appareo) with comparison to colonoscopy | Through study completion, an average of 6 months
  A diagnostic colonoscopy procedure is the reference method. Lesions will be confirmed as malignant by histopathologic examination. The Reduced representation bisulfite sequencing (RRBS) technology to obtain multidimensional variation information on cell-free DNA (cfDNA) methylation, end sequence, fragment size distribution, and copy number variation in the blood, and integrate analysis through machine learning algorithms to accurately assess the risk of colorectal cancer and advanced adenoma. The tests were processed independently of colonoscopy procedure, which was blind to investigators who perform the multiomics profiling and integrate data analysis.

SECONDARY OUTCOMES:
Sensitivity of the multiomics Colorectal Cancer (CRC) screening test (CRC-Appareo) with comparison to FIT, with respect to advanced adenoma (AA) and CRC | Through study completion, an average of 6 months
  A diagnostic colonoscopy procedure is the reference method. Lesions will be confirmed as malignant by histopathologic examination. The the multiomics Colorectal Cancer (CRC) screening test (CRC-Appareo) and FIT test were performed on the blood and stool sample of the same patient.

CONTACTS AND LOCATIONS:
Overall Officials: sheng dai, MD&PhD, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No